CLINICAL TRIAL: NCT03838029
Title: Perioperative Use of a Beta-adrenergic Blocker and a COX-2 Inhibitor in Patients Undergoing Surgery With Primary Pancreatic Cancer: Intervention Aiming to Reduce Pro-metastatic Processes
Brief Title: Perioperative Intervention to Reduce Metastatic Processes in Pancreatic Cancer Patients Undergoing Curative Surgery
Acronym: BC-PC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0308-17-ASF; MOH_2018-03-12_002226 (Registry Identifier: The Israeli Ministry of Health)
Record Dates: First submitted 2019-01-23; First posted 2019-02-12 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Neoplasms
Keywords: Beta-blocker; Propranolol; COX-2 inhibitor; Etodolac
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Propranolol; Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol and etodolac (Active Comparator): Both study medications will be given orally for an intervention phase of 35 days as follows. Etodolac:400mg PO bid for the entire intervention period,Propranolol:20 mg PO bid for 5 preoperative days, 80 mg PO bid on the day of surgery and the following morning, 40 mg PO bid for following 6.5 days, and 20 mg PO bid for next 22 days.
  Interventions: Drug: Propranolol and etodolac
- Placebo (Placebo Comparator): Same schedule as in the active comparator arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propranolol and etodolac — A perioperative combined drug regimen
  Other Names: Deralin and etopan
  Arms: Propranolol and etodolac
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In Israel, of the ~1000 patients diagnosed annually with pancreatic cancer (PC), approximately 250 (25 percent) will be eligible for curative surgery, of which 80 percent will succumb to post-surgical metastatic disease. A reduction in post-surgical metastatic disease will save dozens of patients in Israel annually, and tens-of thousands-around the world. The short perioperative period (days to weeks around surgery) is characterized by stress-inflammatory responses, including catecholamines (CAs, e.g., adrenaline) and prostaglandins (PGs, e.g., prostaglandin-E2) release, and induce deleterious pro-metastatic effects. Animal studies implicated excess perioperative release of CAs and PGs in facilitating cancer progression by affecting the malignant tissue, its local environment, and anti-metastatic immune functions. Congruently, our animal studies indicate that combined use of the beta-adrenergic blocker, propranolol, and the prostaglandins inhibitor, etodolac - but neither drug separately - efficiently prevented post-operative metastatic development. We recently conducted two clinical trials in three medical centers in Israel, recruiting breast (n=38) and colorectal (n=34) cancer patients, assessing the safety and short-term efficacy of perioperative propranolol and etodolac treatment. Drugs were well tolerated, without severe adverse events. Importantly, molecular/biological analyses of the excised primary tumor indicated that drug treatment caused promising anti-metastatic transformations, as well as improvements in immune and inflammatory indices. These included (i) decreased tumor cell capacity to migrate, (ii) reduced pro-metastatic capacity of the malignant tissue, and (iii) improvement in immune infiltrating into the tumor (Paper published in Clinical Cancer Research, 2017). Herein, we propose to conduct a double-blind placebo-controlled two-arm Phase II clinical trial in 210 pancreatic cancer patients undergoing curative surgery in Israel. A perioperative 35-day drug treatment will be initiated 5 days before surgery. Primary outcomes will include (i) 1-year disease-free-survival (DFS), and 5-year overall survival (OS); and (ii) biological markers in blood samples, and in the excised tumor tissue. Secondary outcomes will include safety indices and psychological measures of depression, anxiety, distress, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Stage I or II adenocarcinoma of the head, neck, or uncinated- process of the pancreas.
* Surgically resectable disease (R0 or R1) by spiral CT chest and abdomen scan, No distant metastases
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Signed informed consent form
* Willing and able to comply with study procedures
* Men and women from age 20 up to age 80

Exclusion Criteria:

* Patients with metastatic disease, known prior to surgery
* Patients with history or concomitant malignant disease of any type (except for the current pancreatic cancer
* Patients who were treated with chemotherapy in the last 10 years for any reason
* Patients in whom surgical resection is planned without curative intent
* Patients exhibiting levels Carbohydrate antigen (CA) 19-9 above 500
* Patients with renal failure, measured by creatinine level >1.5
* Patients with significant heart failure (NYHA functional class 3 or higher),
* Patients with significant liver failure (known cirrhosis)
* Patients suffering from active asthma
* Patients with known allergy to any medication from the non-steroidal anti- inflammatory or beta-blockers drug group
* Patients treated chronically with any type of a beta-adrenergic blocker or a cyclooxygenase (COX) inhibitor
* Patients with bradycardia or second or third degree atrioventricular block (AV) block
* Patients with a history of cerebrovascular accident (CVA) or established diagnosed transient ischemic attack (TIA)
* Patients with prinzmetal's angina
* Patients with right sided heart failure owing to pulmonary hypertension
* Patients with significant diagnosed cardiomegaly
* Patients with (current) pheochromocytoma
* Patients with chronic Digoxin treatment
* Patients with active peptic disease
* Patients with peripheral vascular disease
* Pregnant woman
* Special population with impaired judgment
* Patients currently actively participating in any other clinical trial
* contraindication for Whipple procedure
* Patients suffering from sick sinus syndrome
* Patients with borderline resectable tumors, as defined by one of the following:

  * an infiltration >180° of the portal vein
  * abutment of the tumor to the superior mesenteric artery
  * infiltration of the superior mesenteric artery or the celiac trunk

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-11-20 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of cancer recurrence | From the date of surgery until malignant disease is identified, assessed up to 60 months post-surgery
  Data regrading post-surgical recurrence will be recorded at 1,3,6,12,18,24,36,48, and 60 following surgery
Biomarkers in extracted tumor tissue samples | An average of one year following surgery
  Epithelial-to-mesenchymal-transition ( EMT) status and natural-killer cell, macrophage, T-cell, and B-cell infiltration levels into tumor tissue (as assessed by messenger RNA profiling of tissue samples.
Biomarkers in blood samples | An average of one year following surgery
  Cytokine levels in blood samples (interleukin-6, interleukin-10, C-reactive protein, interferon-gamma, and vascular endothelial growth factor and additional exploratory analysis of other cytokines)

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events | 30 days following surgery
  According to the Clavien-Dindo classification system (7 grades of events depicting the severity of the event)
Depression, Anxiety, Global distress | At baseline and at 30 days post-surgery
  Assessed by changes on the brief symptom inventory 18 questionnaire (this questionnaire assess all three scales for depression, anxiety and global distress)
Fatigue | At baseline and at 30 days post-surgery
  4 items related to fatigue in the 36 item short-form survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Oded Zmora, MD, Principal Investigator — Asaf Harofeh Medical Center
Locations (3):
- Israel (3):
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Asaf Harofeh Medical Center, Ẕerifin

REFERENCES:
- [Result] Haldar R, Shaashua L, Lavon H, Lyons YA, Zmora O, Sharon E, Birnbaum Y, Allweis T, Sood AK, Barshack I, Cole S, Ben-Eliyahu S. Perioperative inhibition of beta-adrenergic and COX2 signaling in a clinical trial in breast cancer patients improves tumor Ki-67 expression, serum cytokine levels, and PBMCs transcriptome. Brain Behav Immun. 2018 Oct;73:294-309. doi: 10.1016/j.bbi.2018.05.014. Epub 2018 May 22. PMID 29800703
- [Result] Shaashua L, Shabat-Simon M, Haldar R, Matzner P, Zmora O, Shabtai M, Sharon E, Allweis T, Barshack I, Hayman L, Arevalo J, Ma J, Horowitz M, Cole S, Ben-Eliyahu S. Perioperative COX-2 and beta-Adrenergic Blockade Improves Metastatic Biomarkers in Breast Cancer Patients in a Phase-II Randomized Trial. Clin Cancer Res. 2017 Aug 15;23(16):4651-4661. doi: 10.1158/1078-0432.CCR-17-0152. Epub 2017 May 10. PMID 28490464